CLINICAL TRIAL: NCT03817957
Title: Safety and Efficacy of Postoperative i.v. Iron Substitution With Polyglucoferron Compared to Ferric Carboxymaltose and Oral Iron in Patients With Diagnosed Iron Deficiency Who Develop Anaemia Peri- or Postoperatively (IDA II)
Brief Title: Postoperative i.v. Iron Substitution in Patients With Diagnosed Iron Deficiency
Acronym: IDA-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Dr. Frank Behrens (Other)
Collaborators: University Hospital Frankfurt, Department of Anaesthesiology (Unknown); IRON4U (Unknown); University Hospital Frankfurt Institute for Biostatistics & Mathematical Modelling (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Frank Behrens, Sponsor representative, Fraunhofer Institute for Translational Medicine and Pharmacology ITMP
Organization: Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP0916_03
Record Dates: First submitted 2018-11-19; First posted 2019-01-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Iron Deficiency Anemia
Keywords: post surgery anemia treatment,
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: 2:2:1 distribution Polyglucoferron, Ferric Carboxymaltose i.v., or oral iron substitution with Ferrous sulfate. After safety assessment of first 35 patients treated with Polyglucoferron or Ferric Carboxymaltose i.v. respectively, Ferric Carboxymaltose arm will be closed.
  Remaining patients will be distributed in an 2:1 mode to Polyglucoferron or oral iron
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polyglucoferron (Experimental): once intravenously, dosing according to Hb-levels and body weight, 500 - 2000 mg
  Interventions: Drug: Polyglucoferron
- Ferric Carboxymaltose (Active Comparator): Once intravenously (a second administration is allowed), dosing according to Hb-levels and body weight (500 - 2000 mg, max. single dose of 1000 mg)
  Interventions: Drug: Ferric carboxymaltose
- Ferrous sulfate (Active Comparator): capsules, orally, dosing 50 mg - 200 mg (50 mg: 1 capsule in total, 200 mg: 4 capsules in total, taken as 2 capsules twice daily), duration of treatment 28 days
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Polyglucoferron — intravenous administration
  Other Names: Feramyl
  Arms: Polyglucoferron
Drug: Ferric carboxymaltose — intravenous administration
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose
Drug: Ferrous Sulfate — oral administration
  Other Names: Ferro sanol duodenal
  Arms: Ferrous sulfate

SUMMARY:
Iron deficiency anaemia (IDA) in postoperative patients with confirmed preoperative iron deficiency (ID) in a population with planned major surgery who need fast replenishment of iron as judged by the treating physician will be treated with i.v. iron using Polyglucoferron, Ferric Carboxymaltose or oral iron

DETAILED DESCRIPTION:
In this study, patients with confirmed and documented preoperative non-anaemic iron deficiency (diagnosis up to 28 days before surgery in routine pre-surgery monitoring) who develop anaemia within 12 to 72 hours after start of surgery (with additional confirmation at Baseline) and for whom fast replenishment of iron stores is necessary, will be included and substituted within 24h after Screening Visit/V1. Peri- or postoperative anaemia will be assessed as soon as possible but earliest 12 h after surgery. For short term safety analysis iron in urine will be measured in the first urine after the end of i.v. administration in the first 35 patients who are eligible for analysis in each i.v. treatment group. Only those patients are eligible for whom haematuria and/or proteinuria are excluded using dip stick test. The Ferric Carboxymaltose treatment arm will be closed if a sufficient number of patients is included for safety analysis.The study will then be continued for assessment of co-primary efficacy endpoint: The effectiveness of postoperative i.v. iron substitution with Polyglucoferron compared to conventional oral iron substitution with Ferrous sulfate (treatment 28 - 35 days) to normalize Hb-values or to increase Hb-values by at least 1.5 g/dl until visit 4 will be evaluated as well as patient related outcomes, such as the decreased need for allogenic blood transfusions. In addition, the well-being of the patient will be assumed to improve after treatment using the SF36 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Males or female; aged ≥ 18 years
* Patients after major surgery (e.g., orthopaedic/trauma, vascular, visceral, cardiac surgery) with risk of Hb reduction and/or blood loss who develop anaemia defined as haemoglobin of <12 g/dL for female and <13 g/dL for men within 12 to 72 h after start of surgery and with confirmation at Baseline
* Confirmed and documented preoperative iron deficiency defined as S-ferritin <100 ng/mL without anaemia (Hb ≥12 g/dL for female and ≥13 g/dL for male) within 28 days before surgery
* need for fast iron replenishment as judged by the treating physician
* Written informed consent; willing/able to comply with the protocol

Exclusion Criteria:

* Pregnancy in female patients or breastfeeding women
* Female patients not willing to use a safe method of contraception (PEARL index <1) for the full study period
* Severe physical inability, e.g., American society of anesthesiologists (ASA) physical status IV or V
* Patients receiving blood transfusion 24 week prior surgery
* Non-iron deficiency anaemia, e.g., known Vitamin B12 or folate deficiency, haemoglobinopathy, or unexplained anaemia
* Anticipated medical need for erythropoiesis-stimulating agents during the main study period
* Patients with hemodynamic instability due to any ongoing bleeding. Absence of ongoing bleeding will be confirmed determined either by decision of two independent physicians or by removal of drainage, whichever occurs earlier in routine care)
* Patients with any contraindication to the investigational products, e.g.,

  1. known sensitivity to iron or an ingredient of the investigational products
  2. Significant history of systemic allergic reactions
  3. Haemachromatosis, thalassemia or TSAT >50% as indicator of iron overload
  4. Acute or chronic intoxication
  5. Infection (patient on non-prophylactic antibiotics)
  6. Chronic liver disease and/or screening Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) above three times the upper limit of the normal range
* Chronic kidney disease, defined as Glomerular Filtration Rate (GFR) <30 mL/min
* Active uncontrolled immune-mediated diseases such as rheumatoid arthritis or inflammatory bowel disease
* Primary haematologic disease
* Drug or alcohol abuse according to WHO definition
* Potentially unreliable patients, and those judged by the investigator to be unsuitable for the study
* Current or previous participation in another clinical trial during the last 90 days before screening
* Exclusion criteria related to Ferrous sulfate

  1. according to Summary of product characteristics (SmPC)
  2. hypersensitivity to any ingredient in the formulation
  3. concomitant parenteral iron
  4. haemochromatosis, and other iron overload syndromes
* Exclusion criteria related to Ferric Carboxymaltose:

  1. according to Summary of product characteristics (SmPC)
  2. hypersensitivity to the active substance, to Ferric Carboxymaltose or any of its excipients
  3. known serious hypersensitivity to other parenteral iron products
  4. anaemia not attributed to iron deficiency
  5. evidence of iron overload or disturbances in the utilisation of iron
* Exclusion criteria related to Polyglucoferron

  1. hypersensitivity to any ingredient in the formulation
  2. known serious hypersensitivity to other parenteral iron products
  3. anaemia not attributed to iron deficiency
  4. evidence of iron overload or disturbances in the utilisation of iron

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve normalized Hb-levels or increased Hb of at least 1.5 g/dl | Baseline to approximately 30 days post-baseline (visit 4)
  Proportion of patients in the Polyglucoferron i.v. arm compared to oral iron substitution with Ferrous sulfate at visit 4 compared to Baseline (BL)
pre post difference of volumen-corrected urine iron levels | urine sampled prior to administration and approximately 1 to 8 hours post-baseline
  Pre-post difference of volume-corrected urine iron levels measured before and in the first urine after the end of i.v. administration, defined as short term safety surrogate marker after administration of the i.v. treatments, compared between Polyglucoferron and Ferric Carboxymaltose (volume corrected iron urine is defined as the ratio between urine iron and urine creatinine).

SECONDARY OUTCOMES:
Proportion of patients with normalization of Hemoglobin (Hb) at visit 4 | 30 days after baseline (Visit 4)
  measurement of normalization of Hb defined in World Health Organization (WHO) classification
Level of Hb until visit 4 | Baseline to 30 days after baseline (visit 4)
  determination of levels of Hemoglobin (Hb) (comparison to baseline)
Level of Transferrin Saturation (TSAT) until visit 4 | Baseline to 30 days after baseline (visit 4)
  determination of levels of Transferrin Saturation (TSAT) (mean values in comparison to baseline)
Level of serum-iron until visit 4 | Baseline to 30 days after baseline (visit 4)
  determination of levels of serum-iron (mean values in comparison to baseline)
Level of serum-transferrin until visit 4 | Baseline to 30 days after baseline (visit 4)
  determination of levels of serum-transferrin (mean values in comparison to baseline)
Level of serum-ferritin until visit 4 | Baseline to 30 days after baseline (visit 4)
  determination of levels of serum-ferritin (mean values in comparison to baseline)
Value of serum-phosphate levels at visit 4 (i.v. groups only) | baseline and 30 days after baseline (visit 4)
  measurement of serum-phosphate levels (mean values in comparison to baseline)
Overall tolerability and number, incidence, seriousness, severity, relationship of Adverse Events (AE) and serious adverse events (SAE) until 30 days after Investigational medicinal product (IMP) administration | baseline to 30 days after last IMP administration
  determination of number, incidence, seriousness, severity and causality of adverse events and serious adverse events
Level of c-reactive protein on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of C reactive protein (description of changes in values in comparison to baseline)
Values of ALT on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of ALT (description of changes in values in comparison to baseline)
Values of AST on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of AST (description of changes in values in comparison to baseline)
Values of gamma-glutamyltransferase on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of gamma-glutamyltransferase (description of changes in values in comparison to baseline)
Values of urea nitrogen on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of urea nitrogen (description of changes in values in comparison to baseline)
Values of serum creatinine on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of serum creatinine (description of changes in values in comparison to baseline)
Values of white blood cells on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of white blood cells (description of changes in values in comparison to baseline)
Values of thrombocytes on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of values of thrombocytes (description of changes in values in comparison to baseline)
Changes in systolic blood pressure on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of vital signs as systolic blood pressure
Changes in body temperature on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of body temperature
Changes in pulse rate on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of pulse rate
Changes in diastolic blood pressure on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of vital signs as diastolic blood pressure
Assessment of general conditions on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of general condition will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of Skin on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of Skin will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of eyes on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of eyes will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of ears on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of ears will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of mouth on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of mouth will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of nose on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of nose will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of throat on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of throat will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of cardiovascular system on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of cardiovascular system will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of respiratory system on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of respiratory system,will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of abdomen on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of abdomen will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of gastrointestinal tract on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of gastrointestinal tract will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
clinical assessments of kidneys on each available visit | baseline to 30 days after baseline (visit 4)
  Documentation of clinical assessments of kidneys will be made by investigator - changes to preceding visits and in comparison to baseline will be documented
AEs related to injection/ infusion site reactions (i.v. treatment arms only) and hypersensitivity reactions | baseline to 30 days after last IMP administration
  Documentation of numbers of adverse events related to injection/infusion site reactions (i.v. treatment arms only) and hypersensitivity reactions
Number of deaths from any cause until visit 4 | baseline to 30 days after baseline (visit 4)
  documentation of number of deaths
Proportion of units of allogenic red blood cell transfusion from BL until visit 4 | Baseline to 30 days after baseline (visit 4)
  Documentation of number of units of allogenic red blood cell transfusion
Proportion of patients with need of allogenic red blood cell transfusion from BL until visit 4 | Baseline to 30 days after baseline (visit 4)
  Documentation of the use of allogenic red blood cell transfusion
treatment effect on change in Quality of Life (SF36) at visit 4 compared to BL | Baseline to 30 days after baseline (visit 4)
  documentation of quality of life in the Short Form Health Survey (SF36) with 36 items relying upon patient self-reporting. It contains eight sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. The SF-36 consists of eight scaled scores which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Duration of hospital stay (days) until visit 4 | Baseline to 30 days after baseline (visit 4)
  documentation of days in hospital
Level ofl iron in plasma after end of iron administration (for the i.v. groups (safety analysis group) only) | time points directly after administration of intravenous (i.v.) treatment (approximately 15 minutes post-baseline)
  measurement of iron level in plasma
Level of iron in plasma after urine sampling (for the i.v. groups (safety analysis group) only) | time points after urine sampling (approximately 1 to 8 hours post-baseline)
  measurement of iron level in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, MD, Principal Investigator — University Hospital of Goethe-University Frankfurt
Locations (1):
- Department of Anaesthesiology, Intensive Care Medicine and Pain Therapy, University Hospital of Goethe-University, Frankfurt, Hessia, Germany

IPD SHARING:
Plan to Share IPD: No